CLINICAL TRIAL: NCT02125227
Title: A Randomized, Open-label, Single-dose, 2-Way Cross-over Study to Compare the Safety and the Pharmacokinetic Characteristics of the Co-administration of Rosuvastatin and Metformin SR and YH14755 and to Investigate the Effect of Food on the Pharmacokinetics of YH14755
Brief Title: Phase 1 Clinical Trial to Investigate the Effect on the Pharmacokinetics of YH14755 Compared to Co-administration of Rosuvastatin and Metformin SR in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: YH14755-102
Record Dates: First submitted 2014-04-24; First posted 2014-04-29 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Rosuvastatin Calcium; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 of Study A (Experimental): single dosing of Rosuvastatin and Metformin 14 days later, single dosing of YH14755
  Interventions: Drug: Rosuvastatin, Metformin, YH14755
- Group 2 of Study A (Experimental): single dosing of YH14755 14 days later, single dosing of Rosuvastatin and Metformin
  Interventions: Drug: Rosuvastatin, Metformin, YH14755
- Group 1 of Study B (Experimental): single dosing of YH14755 with fasting state 14 days later, single dosing of YH14755 after having breakfast
  Interventions: Drug: YH14755
- Group 2 of Study B (Experimental): single dosing of YH14755 after having breakfast 14 days later, single dosing of YH14755 with fasting state
  Interventions: Drug: YH14755

INTERVENTIONS:
Drug: Rosuvastatin, Metformin, YH14755 — single dose
  Other Names: Crestor, GlucodaunOR, YH14755
  Arms: Group 1 of Study A; Group 2 of Study A
Drug: YH14755 — single dose
  Arms: Group 1 of Study B; Group 2 of Study B

SUMMARY:
The objective of this study is to Compare the Safety and the Pharmacokinetic Characteristics of the Co-administration of Rosuvastatin and Metformin SR and YH14755 and to Investigate the Effect of Food on the Pharmacokinetics of YH14755 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female with a body mass index(BMI) between 18.5 and 25 kg/m2
2. Who has not suffered from clinically significant disease
3. Provision of signed written informed consent

Exclusion Criteria:

1. History of and clinically significant disease
2. A history of drug abuse or the presence of positive reactions to drugs that have abuse potential in urine screenings for drugs.
3. Administration of other investigational products within 3 months prior to the first dosing.
4. Administration of herbal medicine within 4 weeks or administration of ethical drugs within 2 weeks or administration of over-the-counter (OTC) drugs within 1 week prior to the first dosing of the investigational product (if the investigator (study doctor) determines that the person meets other criteria appropriately, the relevant person may participate in the study).
5. Volunteers considered not eligible for the clinical trial by the investigator (study doctor) due to reasons including laboratory test results, ECGs, or vital signs.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
AUClast of rosuvastatin and metformin | 0~48hr, totally 17 points
Cmax of rosuvastatin and metformin | 0~48hr, totally 17 points

SECONDARY OUTCOMES:
Tmax of rosuvastatin and metformin | 0~48hr, totally 17 points
t1/2 of rosuvastatin and metformin | 0~48hr, totally 17 points
%AUC of rosuvastatin and metformin | 0~48hr, totally 17 points
AUCinf of rosuvastatin and metformin | 0~48hr, totally 17 points

CONTACTS AND LOCATIONS:
Overall Officials: Mingul Kim, MD, Ph.D, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea